CLINICAL TRIAL: NCT00541892
Title: Sibling Oocyte Study of Medium for IVF/ICSI With no Human Serum Albumine
Brief Title: Sibling Oocyte Study of Medium for In Vitro Fertilization/Intracytoplasmic Sperm Injection (IVF/ICSI) With no Human Serum Albumine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: senior coworker retired
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Cellcura AS (Industry); Vekst i Grenland (Unknown); Innovation Norway (Unknown)
Responsible Party: Principal Investigator, Hans Ivar Hanevik, PhD, Sykehuset Telemark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s-05249; 14231(NSD)
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: In Vitro Fertilization; Infertility
Keywords: Cell Culture Techniques
MeSH Terms: conditions — Infertility | interventions — Culture Media

ARMS (2):
- 1 (Experimental): Medium with no human serum albumine added
  Interventions: Other: Medium with no human serum albumine added
- 2 (Active Comparator): Conventional medium
  Interventions: Other: Conventional medium

INTERVENTIONS:
Other: Medium with no human serum albumine added — See above
  Arms: 1
Other: Conventional medium — See above
  Arms: 2

SUMMARY:
The purpose of this study is to determine if a new medium with no human serum albumine added is as good as the media conventionally used for IVF/ICSI.

DETAILED DESCRIPTION:
Cells attained in IVF/ICSI procedures are kept in a medium that nurture the cells. Until now all such media have contained human serum albumine. The purpose of this study is to determine if a new medium with no human serum albumine added is as good as the media conventionally used for IVF/ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Couples seeking IVF/ICSI.
* Female under 38 years of age.
* No more than two previous IVF/ICSI treatments without pregnancy.
* Regular menstruation periods.
* No endocrine disease that requires treatment in the female.
* BMI below 30 in the female.
* At least 8 mature follicles upon monitoring or 6 MII oocytes upon ICSI.
* Written informed consent.

Exclusion Criteria:

* Low responders to FSH.
* Females in danger of developing OHSS.
* Sperm sample below ICSI-quality.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Fertilization | 24 hours
Cleavage | 48 hours
Embryo score | 48 hours
Embryos used | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jarl Kahn, Dr. Med, Study Director — Fertilitetsklinikken Sør
Locations (1):
- Fertilitetsklinikken Sør, Porsgrunn, Telemark, Norway